CLINICAL TRIAL: NCT02964897
Title: Veterans Justice Reentry (Post-Incarceration) (QUE 15-284)
Brief Title: Improving Linkage to Health and Other Services for Veterans Leaving Incarceration
Acronym: PIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: QUX 16-012; QUE 15-284 (Other Grant/Funding Number: HSR&D QUERI)
Record Dates: First submitted 2016-11-04; First posted 2016-11-16 (Estimated); Results first posted 2021-10-08 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Linkage to Care; Homelessness; Substance Use Disorder; Mental Health
Keywords: justice involvement; Homeless; Vulnerable Populations; Linkage to care; Veterans
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm with Peer Support (Experimental): Veterans in this arm will receive the peer-support intervention, in addition to the usual care from the Health Care for Reentry Veterans Program.
  Interventions: Behavioral: Peer-support plus usual care from the Health Care for Reentry Veterans program
- Comparison Arm with Usual Care (Other): Veterans in this arm will be receiving usual care from the Health Care for Reentry Veterans program (but they will not receive the peer-support intervention). They will be selected to be frequency-matched to veterans in the intervention arm by date of release from incarceration.
  Interventions: Behavioral: Usual care from the Health Care for Reentry Veterans program

INTERVENTIONS:
Behavioral: Peer-support plus usual care from the Health Care for Reentry Veterans program — a peer mentor who is also a veteran will establish a relationship with each subject and provide instrumental and emotional support to the subject during the first 6 months of the subject's release from incarceration. This is in addition to the usual reentry support provided by the Health Care for Reentry Veterans program.
  Other Names: peer mentoring; forensic peer support
  Arms: Intervention Arm with Peer Support
Behavioral: Usual care from the Health Care for Reentry Veterans program — Health Care for Reentry Veterans program provides reentry planning while the veteran is incarcerated. An outreach worker visits the veteran in the incarceration facility to conduct a needs assessment and help create a reentry plan to cover issues such as where they will be housed, what health care appointments they will need in the first 30 days, whether they need legal assistance, etc.
  Other Names: HCRV reentry support
  Arms: Comparison Arm with Usual Care

SUMMARY:
Veterans leaving incarceration and re-entering their communities (often described as "reentry" Veterans) face a number of challenges, including uncertainty about housing, vulnerability to substance use and relapse, on-going mental health concerns, and often multiple health conditions require timely continuity of care. The purpose of the project is to increase support for Veterans post-incarceration through the addition of trained peers with lived experience of being a Veteran and a history of incarceration. Emphasis will be on peers who will help link Veterans to Veterans Health Administration (VHA) services, including housing and healthcare. Peers will provide linkage with Health Care Reentry Veterans program specialists, transportation to appointments, and support in community reintegration. Peers will assist reentry veterans to make a successful transition and get and stay engaged in their care.

DETAILED DESCRIPTION:
Veterans leaving incarceration (henceforth, "reentry Veterans") are among the most underserved by the VA and thus are an increasingly high priority population. The Bureau of Justice Statistics estimates that 140,000 Veterans are incarcerated in the U.S. at a given time, approximately 80% of whom are eligible for VA benefits. Many of these Veterans had problems with substance use disorders (SUD)(including alcohol) and/or mental health (MH) issues prior to being incarcerated.

The VA's national Health Care for Reentry Veterans (HCRV) program identifies 10,000-15,000 incarcerated Veterans annually preparing to transition back to the community. A HCRV outreach specialist works with incarcerated VHA-eligible Veterans to establish a post-release plan for linkage to VHA services. This program, with 1-2 outreach specialists per state, has improved the connection between reentry Veterans and the VHA. However, the investigators' analyses of homeless program data linked to VHA administrative data indicate that 43% of eligible HCRV Veterans do not have a VHA outpatient contact in the first 4 months post incarceration. Reducing this number is critical given the elevated rates of chronic health conditions, as well as MH or SUDs in this population.

To address this gap, the investigators will work with the national HCRV office to implement an evidence-based peer support intervention to extend the reach and effectiveness of the HCRV program in linking Veterans to VHA. Peers with incarceration experience are likely to better understand and connect with Veterans on a personal level than the outreach specialist, and thus are more likely to maintain contact and link to VHA during the first months post-release. Peers are gaining popularity in forensic settings (called "forensic peer specialists") with civilian populations and would likely be beneficial for a Veteran population .

The aims of this project are:

1. Conduct contextual analysis to identify VHA and community reentry resources, and to describe how reentry Veterans use them.
2. Implement peer-support, in one state, to link reentry veterans to VHA primary, mental health, and SUD services. The investigators will use external and internal facilitation as the implementation strategy.
3. Spread the peer-support intervention to another, geographically, and contextually different state.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* Veteran released from a Massachusetts state prison or county jail.
* (for intervention subjects: interested in receiving reentry services) Phase 2
* Veteran released from a Connecticut state prison or jail.
* (for intervention subjects: interested in receiving reentry services)

Exclusion Criteria:

- No history of dementia or other serious cognitive condition that would prevent them from being interviewed or completing a survey questionnaire.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald K McInnes, ScD MS BA, Principal Investigator — VA Bedford HealthCare System, Bedford, MA; Allen L. Gifford, MD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim B, McCullough MB, Simmons MM, Bolton RE, Hyde J, Drainoni ML, Fincke BG, McInnes DK. A novel application of process mapping in a criminal justice setting to examine implementation of peer support for veterans leaving incarceration. Health Justice. 2019 Mar 26;7(1):3. doi: 10.1186/s40352-019-0085-x. PMID 30915620
- [Derived] Simmons MM, Fincke BG, Drainoni ML, Kim B, Byrne T, Smelson D, Casey K, Ellison ML, Visher C, Blue-Howells J, McInnes DK. A two-state comparative implementation of peer-support intervention to link veterans to health-related services after incarceration: a study protocol. BMC Health Serv Res. 2017 Sep 12;17(1):647. doi: 10.1186/s12913-017-2572-x. PMID 28899394

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm With Peer Support | Comparison Arm With Usual Care
Started | 43 | 36
Completed | 43 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm With Peer Support | Comparison Arm With Usual Care | Total
Number analyzed (Participants) | 43 | 36 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (13) | 53.8 (14) | 51.4 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 43 | 36 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American or Black | 10 | 6 | 16
  Race: White | 31 | 30 | 61
  Race: Multiple/other/declined | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 36 | 79
Marital status [Count of Participants; unit: Participants]
  Not partnered (single, divorced, separated, widowed) | 37 | 34 | 71
  Married or other partner relationship | 6 | 2 | 8
Self-rated health [Count of Participants; unit: Participants]
  Excellent | 6 | 8 | 14
  Very good | 9 | 3 | 12
  Good | 17 | 12 | 29
  Fair | 8 | 5 | 13
  Poor | 3 | 4 | 7
  Missing | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Substance Use Care
Description: Participant will have made and kept one or more substance use disorder care visits
Time Frame: 3 months after release from incarceration
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm With Peer Support | Comparison Arm With Usual Care
Number analyzed (Participants) | 43 | 36
Participants | 37 | 7

2. Primary Outcome: Mental Health
Description: Participant will have made and kept one or more outpatient mental health care visits
Time Frame: 3 months after release from incarceration
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm With Peer Support | Comparison Arm With Usual Care
Number analyzed (Participants) | 43 | 36
Participants | 42 | 23

3. Primary Outcome: Primary Care
Description: Participant will have made and kept one or more primary care visits
Time Frame: 3 months after release from incarceration
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm With Peer Support | Comparison Arm With Usual Care
Number analyzed (Participants) | 43 | 36
Participants | 25 | 24

ADVERSE EVENTS:
Time Frame: 1 Year
Description: For the comparison group it was a historical control, only those living were included.
Arm/Group | Intervention Arm With Peer Support | Comparison Arm With Usual Care
All-Cause Mortality (participants affected / at risk) | 1/43 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/36
Other Adverse Events (participants affected / at risk) | 0/43 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm With Peer Support (N=43) | Comparison Arm With Usual Care (N=36)
Death (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Because of our use of a historical comparison group, the context in which they received reentry services and their individual characteristics may have differed from the intervention group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT02964897/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT02964897/SAP_001.pdf